CLINICAL TRIAL: NCT03527225
Title: A Randomized Trial of Music to Decrease Anxiety in Women Starting Radiation Therapy for Cancer
Brief Title: Music of Choice to Decrease Anxiety During Radiation Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201703352; OCR17059 (Other: Office of Clinical Research)
Record Dates: First submitted 2018-05-04; First posted 2018-05-17 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Anxiety; Cancer
Keywords: Music Therapy; First Radiotherapy; Anxiety Reduction; Psychosocial Functioning; State - Trait Anxiety Inventory (STAI); Symptom Distress Thermometer (SDT)
MeSH Terms: conditions — Anxiety Disorders; Neoplasms | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Consented, eligible female subjects to be randomized to "Music" or "No Music" to evaluate pre and post treatment anxiety level via STAI and SDT anxiety questionnaire at their first radiotherapy treatment for cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music (Experimental): Patients randomized to the music intervention arm will select a preferred genre of music from an internet based resource.
  Interventions: Other: Music
- No Music (No Intervention): These patient's will have no music playing during the first radiotherapy session.

INTERVENTIONS:
Other: Music — The patient's preferred music will be played during the first radiotherapy treatment session from speakers located inside the treatment room. The duration of the music will be 10 to 20 minutes. The music will be turned off at the patient's request if it bothers them. Length of music playing and if the patient requested that it be turned off, will be recorded.
  Arms: Music

SUMMARY:
The primary hypothesis of the study is that listening to music will reduce anxiety in female cancer patients during the first radiotherapy treatment session.

DETAILED DESCRIPTION:
Receiving radiotherapy induces anxiety in at least 1/3 of patients who did not have a previously existing anxiety condition1. Female gender is a positive predictive factor for psychosocial decline during radiotherapy. One-fourth of patients disrupt their planned radiotherapy treatment course due to anxiety. Music therapy has demonstrated effectiveness in reducing anxiety when implemented in other medical settings including mechanical ventilation, burn debridement and venipuncture in pediatric patients. There have been some trials which have found a reduction in anxiety when pre-recorded music along with other relaxation techniques have been implemented during radiotherapy. This trial seeks to investigate the benefit of pre-recorded music alone in reducing anxiety experienced during the first radiotherapy treatment session in female cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to receive radiotherapy for malignant tumor
* ECOG Performance Status 0-4
* Fluent in English Language
* Inclusion in this study will not be based on race or ethnicity
* Patients must be deemed able to comply with the treatment plan.
* Patients must provide study specific informed consent prior to study entry.

Exclusion Criteria:

* Prior history of radiation therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Multiple studies document a higher rate of psychological distress in female cancer patients.The study is limited to females to decrease confounding prognostic factors related to anxiety during cancer therapy. By restricting enrollment to women in this study, is to gain proof of concept that the intervention is effective and can be determined with a smaller sample size.
Enrollment: 135 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Mean change of STAI Score from within 2 hours prior to first RT session to 2 hours post first RT session. | baseline
  Percent change in mean anxiety score as measured with the State-Trait Anxiety Inventory (STAI) questionnaire. Assessed by the mean value (pre minus post radiotherapy STAI score) divided by mean pre-treatment score multiplied by 100. A score of 39-40 on each subset suggests clinically significant anxiety.

SECONDARY OUTCOMES:
Mean change of SDT Score from within 2 hours prior to first RT session to 2 hours post first RT session. | baseline
  Percentage change in mean anxiety score as measured with the Symptom Distress Thermometer (SDT). Scale of 0 - 10; with 10 being clinically significant distress.
Magnitude change of STAI Score | baseline
  The magnitude of change in anxiety score of STAI in "high anxiety" patients (pre-treatment STAI ≥ 40) as a result of listening to music during the first radiotherapy session.
Magnitude change of SDT Score from within 2 hours prior to first RT session to 2 hours post first RT session. | baseline
  The magnitude of change in anxiety score of SDT in "high anxiety" patients (pre-treatment SDT ≥ 4) as a result of listening to music during the first radiotherapy session. Scale of 0 - 10; with 10 being clinically significant distress.
STAI "High to Low Score" Change from within 2 hours prior to first RT session to 2 hours post first RT session. | baseline
  The number and percentage of patients who drop from a "high" to "low" anxiety level in both intervention groups using STAI scores. A score of 39-40 on each subset suggests clinically significant anxiety.
SDT "High to Low Score" Change from within 2 hours prior to first RT session to 2 hours post first RT session. | baseline
  The number and percentage of patients who drop from a "high" to "low" anxiety level in both intervention groups using SDT scores. Scale of 0 - 10; with 10 being clinically significant distress.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie A. Lockney, M.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida Health Cancer Center, Gainesville, Florida, United States